CLINICAL TRIAL: NCT05961618
Title: Cortical Excitability and Neuropsychological Behavior Changes Following COVID-19 Infection in the Human Brain
Brief Title: Brain Function Changes Following COVID-19 Infection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LY2023-133
Record Dates: First submitted 2023-07-24; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
Keywords: covid-19; TMS; response inhibition; decision-
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Uninfected: Subjects who had recovered from SARS-CoV-2 infection
- Infected: Subjects who had not been infected with SARS-CoV-2.

SUMMARY:
The global COVID-19 pandemic has now led to millions of infections worldwide. It produces long-lasting changes in the general physiology of multiple organs, including the brain. Thus, this study aimed to comprehensively understand the cortical excitability and neuropsychological behavior changes in patients following SARS-CoV-2.

DETAILED DESCRIPTION:
The global COVID-19 pandemic caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) has led to millions of infections and deaths worldwide. However, many issues about the nature of some long-term infection-related symptoms have not yet been well clarified.

Several lines of evidence have shown that SARS-CoV-2 can attack multiple organs such as the lungs, heart, kidneys, liver, as well as brain. The pathophysiologic analyses have shown the impact of SARS-CoV-2 on the brain, including the virus-induced neuroinflammation, the immune reactions, and the possible presence of the coronavirus in the central nervous system in the COVID-19 cases. Indeed, patients who recovered from COVID-19 may experience several long-term symptoms related to brain health, such as fatigue, cognitive and attention deficits, anxiety, and depression, which can affect their ability to work or even daily life. Therefore, the neuropsychological behavior changes in patients following SARS-CoV-2 infection remain an ongoing study area.

In parallel, studies have shown that behavioral abnormities in COVID-19 patients are often accompanied by cortical changes. Utilizing magnetic resonance imaging, a more significant reduction in grey matter thickness and tissue contrast in the orbitofrontal cortex and parahippocampal gyrus has been identified. Other studies confirmed impairment of frontoparietal cognitive functions and frontoparietal hypometabolism by 18F-fluoro-2-deoxy-d-glucose positron emission tomography15. In addition, electroencephalogram abnormalities were also seen in patients who survived from COVID-19. In recent decades, transcranial magnetic stimulation (TMS) has been recognized as a promising and noninvasive adjuvant diagnostic tool enabling assessment of the excitatory and inhibitory properties of the motor cortex as well as brain connectivity17,18. However, the evidence of inhibitory or excitatory changes of intracortical networks in patients recovered from COVID-19 is still scarce.

In this study, we aimed to investigate whether deficits in response inhibition and decision-making could be found in patients following mild SARS-CoV-2 infection. Moreover, we also focused on the neurophysiological evaluation of excitability and neurotransmission within the primary motor cortex (M1).

ELIGIBILITY:
Inclusion Criteria:

* 1. Age between 18 and 60 years; 2. Completed the TMS and cognitive function tests; 3. Without physical discomfort or special physiological conditions (e.g., female subjects in their menstrual cycle or ovulation)

Exclusion Criteria:

* 1. Had previous history of neurological or psychiatric disorders; 2. Had cognitive impairment or use of recreational or therapeutic psychoactive drugs within the past three months;3. Had severe hepatic or renal impairment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The medical record of subjects who received cognitive function and TMS tests between January 2023 and March 2023 by our investigation group were retrospectively analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
The cortical excitability changes following COVID-19 infection. | January 2023 to March 2023
  This was assessed by single/paired pulse TMS procedures.

SECONDARY OUTCOMES:
The neuropsychological behaviors following COVID-19 infection. | January 2023 to March 2023
  These were assessed by Stop-signal task (SST) and Choice under risk and ambiguity task (CRA).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang Y, Yang H, Wang C, Yuan TF, Zhang S. Reduced risk tolerance and cortical excitability following COVID-19 infection. CNS Neurosci Ther. 2024 Aug;30(8):e14879. doi: 10.1111/cns.14879. No abstract available. PMID 39107954